CLINICAL TRIAL: NCT06215053
Title: The Effect of Erector Spinal Area (Esp) Block Applied Before or After Surgery on Postoperative Acute Pain and Quality of Recovery in Patients Undergoing Spinal Surgery
Brief Title: Pre-post Erector Spine Plane Block-spinal Surgery
Acronym: pre-post-esp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, anesthesiologist, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 21-12-2023
Record Dates: First submitted 2023-12-21; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use; Pain, Acute
Keywords: erector spinae block; postoperative pain; spinal surgery
MeSH Terms: conditions — Acute Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized double blinding
Who Masked: Participant, Care Provider
Masking Description: Blind patients and postoperative follow-ups will not know which group the patient is in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Other): Following induction of anesthesia, ESP block will be performed before the surgery begins
  Interventions: Other: erector spine plane block
- group 2 (Other): An ESP block will be performed before waking the patient at the end of surgery.
  Interventions: Other: erector spine plane block

INTERVENTIONS:
Other: erector spine plane block — After anesthesia and surgical procedures, bilateral ESP block will be applied under ultrasonography guidance from the midline 3 cm lateral from the T10 level. After cleaning the area with povidone-iodine before the block, the T10 transverse protrusion will be determined using a linear ultrasound probe. Local anesthetic will be applied between the transverse process and the erector spinae muscle with the help of an insulated needle designed for peripheral block procedures. The location of the needle will be confirmed by hydrodissection with physiological saline without local anesthesia. After the location of the needle is confirmed, 20 ml of LA and saline mixture will be applied and the same process will be repeated in the contralateral side. Of the total 40 ml LA, 20 ml will consist of bupivacaine 0.5% (MARCAİNE), 10 ml will consist of lidocaine 2% (Aritmal), and 10 ml will consist of physiological saline.
  Other Names: esp block

SUMMARY:
Spinal surgery patients generally have chronic pain in the preoperative period and are exposed to widespread and severe acute pain postoperatively. In spinal surgery patients, providing postoperative analgesia is important not only for the patient's comfort but also for preventing the negative effects of pain on the systems, allowing early mobilization, reducing hospital stay and especially reducing chronic pain syndrome.

Although ESP block is routinely used in spinal analgesia, the answer to the question of whether investigators should perform the block after putting the patient to sleep or before waking the patient after completing the surgery is not clear. Preference varies among anesthesiologists.YOU investigators propose a randomized double-blind study comparing patients who underwent ESP block before surgery (Group 1) with patients who underwent ESP block after surgery (Group 2).

DETAILED DESCRIPTION:
investigators propose a randomized double-blind study comparing patients who underwent ESP block before surgery (Group 1) with patients who underwent ESP block after surgery (Group 2). Blind patients and postoperative follow-ups will not know which group the patient is in the study. The study will be conducted at Adnan Menderes University hospital with the approval of the ethics committee and the written consent of the patients. The study will be registered on the ClinicalTrials.gov website before the first patient is enrolled.

Preoperative Visit Documentation of eligibility and consent will be confirmed at the preoperative visit. During this visit, patients will provide demographic and historical medical information, including information regarding medication use. They will fill out the QR-40 quality compilation survey form.

intraoperative The clinic's routine anesthesia protocol will be applied to the patient. Anesthesia will not be interfered with.

Group 1: Following induction of anesthesia, ESP block will be performed before the surgery begins, Group 2: ESP block will be performed before waking the patient at the end of surgery.

Postoperative The peroperative analgesia plan will be applied the same to all patients. In this protocol, intravenous paracetamol was determined as 1 g and tramadol was determined as 1 mg/kg. Then it is paracetamol every eight hours and tramadol from PCA.

At the end of the operation, patients' pain levels will be determined and recorded with the Numeric Rating Scale (NRS) system at postoperative intervals.

The quality of recovery (QoR-40) of both groups of patients at the 24th postoperative hour will be evaluated with a scoring system.

ELIGIBILITY:
Inclusion Criteria:

1. Spinal surgery performed under elective conditions
2. ASA I-III 3.18-75 years old

Exclusion Criteria:

1. Rejection during registration
2. Request for dismissal from employment
3. Inability to give informed consent
4. Emergency surgery
5. Bleeding diathesis
6. Presence of contraindications to the LA agents used in this study
7. Chronic use of opioids
8. Psychiatric disorders
9. Presence of infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
opioi consumption | 24 hours
  Postoperative 30th minute, 1st, 6th, 12th, 18th. Patients' opioid consumption on the PCA will be recorded at the 24th and 24th hours.

SECONDARY OUTCOMES:
nrs | 24 hours
  Preoperative period and Postoperative 30th minute, 1st, 6th, 12th, 18th. And at the 24th hour, patients' pain levels and NRS scores will be recorded.

OTHER OUTCOMES:
recovery | 24 hours
  The quality of recovery of patients at the preoperative and postoperative 24th hour will be evaluated with a scoring system (QoR-40).The QoR-40 is a recovery-specific and patient-rated questionnaire that contains 40 items measuring five dimensions: the physical comfort (12 items), emotional state (nine items), physical independence (five items), psychological support (seven items) and pain (seven items).The total score and subscales of the QoR-40 are measured using a five-point Likert scale (for positive items: 1 = none of the time, 5 = all of the time; for negative items, the scoring was reversed) and individual scores are then added together, with the minimum score being 40 points and the maximum score being 200 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Ferdi Gülaştı, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No